CLINICAL TRIAL: NCT05139810
Title: A Phase 3 Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of ISIS 721744 in Patients With Hereditary Angioedema (HAE)
Brief Title: OASIS-HAE: A Study to Evaluate the Safety and Efficacy of Donidalorsen (ISIS 721744 or IONIS-PKK-LRx) in Participants With Hereditary Angioedema (HAE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISIS 721744-CS5; 2021-002571-19 (EudraCT Number)
Expanded Access: NCT06415448 (Available)
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Hereditary Angioedema
Keywords: HAE
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — donidalorsen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pooled Placebo (Placebo Comparator): Participants with hereditary angioedema type I/type II (HAE-1/HAE-2) received placebo subcutaneously (SC) either every 4 weeks (Weeks 1, 5, 9, 13, 17, and 21) or 8 weeks (Weeks 1, 9, and 17)
  Interventions: Drug: Donidalorsen
- Cohort A: Donidalorsen 80 mg (Experimental): Participants with HAE-1/HAE-2 received donidalorsen, 80 mg, SC, every 4 weeks at Weeks 1, 5, 9, 13, 17, and 21.
  Interventions: Drug: Donidalorsen
- Cohort B: Donidalorsen 80 mg (Experimental): Participants with HAE-1/HAE-2 received donidalorsen, 80 mg, SC, every 8 weeks at Weeks 1, 9, and 17.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donidalorsen — Donidalorsen was administered by SC injection.
  Arms: Cohort A: Donidalorsen 80 mg; Pooled Placebo
Drug: Placebo — Donidalorsen-matching placebo was administered by SC injection.
  Arms: Cohort B: Donidalorsen 80 mg

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of donidalorsen in participants with HAE and effect of donidalorsen on the quality and pattern of HAE attacks and their impact on quality of life (QoL).

DETAILED DESCRIPTION:
This was a Phase 3, multi-center, double-blind, randomized, placebo-controlled study of donidalorsen in 91 participants. Participants were randomly assigned in a 2:1 ratio to Cohort A (donidalorsen or placebo every 4 weeks) or Cohort B (donidalorsen or placebo every 8 weeks), respectively. Within each Cohort, participants were randomized in a 3:1 ratio to receive donidalorsen or matching-placebo. The study included an up to 8-week Screening Period, a 24-week Treatment Period, and an up to 13-week Post-treatment Period.

ELIGIBILITY:
Key Inclusion Criteria

1. Participants, or their legally appointed and authorized representatives, must provide written and signed informed consent form (ICF)/assent
2. Participants must be aged ≥ 12 years at the time of informed consent and, as applicable, assent
3. Participants must have a documented diagnosis of hereditary angioedema type 1 (HAE-1)/hereditary angioedema type 2 (HAE-2)
4. Participants must:

   1. Experience a minimum of 2 HAE attacks (confirmed by the Investigator) during the Screening Period
   2. Be willing to complete the participant reported outcomes (PRO) assessments throughout the study
5. Participants must have access to, and the ability to use acute medication(s) to treat angioedema attacks

Key Exclusion Criteria

1. Concurrent diagnosis of any other type of recurrent angioedema, including acquired, idiopathic angioedema or HAE with normal C1-INH (also known as HAE Type III)
2. Any clinically-significant abnormalities in screening laboratory values that would render a participant unsuitable for inclusion in the study
3. Treatment with another investigational drug or biological agent within 1 month or 5 half-lives, whichever is longer, of Screening
4. Participated in a prior ISIS 721744 study
5. Exposure to any of the following medications:

   1. Angiotensin-converting enzyme (ACE) inhibitors or any estrogen containing medications with systemic absorption within 4 weeks prior to Screening
   2. Chronic prophylaxis with Takhzyro, Haegarda, Cinryze and Ruconest or Orladeyo within 5 half-lives prior to Screening
   3. Oligonucleotides (including small interfering ribonucleic acid [siRNA]) within 4 months of Screening if single dose received, or within 12 months of Screening if multiple doses received. This exclusion does not apply to vaccines
6. Recent history (3 years) of, or current drug or alcohol abuse

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (15):
  - Ionis Investigative Site, Scottsdale, Arizona
  - Ionis Investigative Site, San Diego, California
  - Ionis Investigative Site, Santa Monica, California
  - Ionis Investigative Site, Walnut Creek, California
  - Ionis Investigative Site, Colorado Springs, Colorado
  - Ionis Investigative Site, Tampa, Florida
  - Ionis Investigative Site, Kansas City, Kansas
  - Ionis Investigative Site, Boston, Massachusetts
  - Ionis Investigative Site, Ann Arbor, Michigan
  - Ionis Investigative Site, St Louis, Missouri
  - Ionis Investigative Site, Columbus, Ohio
  - Ionis Investigative Site, Toledo, Ohio
  - Ionis Investigative Site, Hershey, Pennsylvania
  - Ionis Investigative Site, Dallas, Texas
  - Ionis Investigative Site, Murray, Utah
- Belgium (2):
  - Ionis Investigative Site, Brussels
  - Ionis Investigative Site, Edegem
- Ionis Investigative Site, Sofia, Bulgaria
- Canada (2):
  - Ionis Investigative Site, Ottawa, Ontario
  - Ionis Investigative Site, Edmonton
- Ionis Investigative Site, Odense, Denmark
- France (3):
  - Ionis Investigative Site, La Tronche
  - Ionis Investigative Site, Marseille
  - Ionis Investigative Site, Paris
- Germany (3):
  - Ionis Investigative Site, Berlin
  - Ionis Investigative Site, Frankfurt
  - Ionis Investigative Site, Munich
- Israel (3):
  - Ionis Investigative Site, Ashkelon
  - Ionis Investigative Site, Haifa
  - Ionis Investigative Site, Tel Aviv
- Italy (5):
  - Ionis Investigative Site, Catania
  - Ionis Investigative Site, Milan
  - Ionis Investigative Site, Napoli
  - Ionis Investigative Site, Padua
  - Ionis Investigative Site, Palermo
- Netherlands (2):
  - Ionis Investigative Site, Amsterdam
  - Ionis Investigative Site, Groningen
- Ionis Investigative Site, Krakow, Poland
- Spain (4):
  - Ionis Investigative Site, Barcelona
  - Ionis Investigative Site, Madrid
  - Ionis Investigative Site, Seville
  - Ionis Investigative Site, Valencia
- Turkey (Türkiye) (3):
  - Ionis Investigative Site, Ankara
  - Ionis Investigative Site, Istanbul
  - Ionis Investigative Site, Izmir
- United Kingdom (3):
  - Ionis Investigative Site, Birmingham
  - Ionis Investigative Site, Bristol
  - Ionis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.
URL: https://vivli.org/ourmember/ionis/

REFERENCES:
- [Result] Riedl MA, Tachdjian R, Lumry WR, Craig T, Karakaya G, Gelincik A, Stobiecki M, Jacobs JS, Gokmen NM, Reshef A, Gompels MM, Manning ME, Bordone L, Newman KB, Treadwell S, Wang S, Yarlas A, Cohn DM; OASIS-HAE Team. Efficacy and Safety of Donidalorsen for Hereditary Angioedema. N Engl J Med. 2024 Jul 4;391(1):21-31. doi: 10.1056/NEJMoa2402478. Epub 2024 May 31. PMID 38819395

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 39 investigative sites from 3 December 2021 to 09 November 2023.
Pre-assignment Details: A total of 91 participants were enrolled and randomized in the study. Out of 91, 1 participant withdrew consent prior to receiving the study drug. As pre-specified in the protocol and statistical analysis plan, for purposes of analysis, data for placebo participants from Cohort A and Cohort B was pooled for comparison to donidalorsen treated participants.
Groups:
- Pooled Placebo: Participants with hereditary angioedema type I/type II (HAE-1/HAE-2) received placebo subcutaneously (SC) either every 4 weeks (Week 1, 5, 9, 13,17, and 21) or 8 weeks (Week 1, 9, and 17).
Period: Overall Study
Arm/Group | Pooled Placebo | Cohort A: Donidalorsen 80 mg | Cohort B: Donidalorsen 80 mg
Started | 22 | 46 | 23
Full Analysis Set (FAS) (The FAS included all randomized participants who received at least 1 dose of the study drug (donidalorsen or placebo).) | 22 | 45 | 23
Completed | 0 | 1 | 3
Not Completed | 22 | 45 | 20
Not completed — Voluntary Withdrawal | 2 | 1 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Roll Over to CS7 | 19 | 44 | 20

BASELINE CHARACTERISTICS:
Population: The FAS included all randomized participants who received at least 1 dose of the study drug (donidalorsen or placebo). As pre-specified in the protocol and statistical analysis plan, for purposes of analysis, data for placebo participants from Cohort A and Cohort B was pooled for comparison to donidalorsen treated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | Cohort A: Donidalorsen 80 mg | Cohort B: Donidalorsen 80 mg | Total
Number analyzed (Participants) | 22 | 45 | 23 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (11.03) | 39.6 (15.23) | 34.1 (13.22) | 37.2 (13.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 28 | 12 | 48
  Male | 14 | 17 | 11 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3 | 6
  Not Hispanic or Latino | 21 | 43 | 20 | 84
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaskan Native | 2 | 0 | 1 | 3
  Race: Asian | 0 | 1 | 0 | 1
  Race: Black or African American | 1 | 1 | 0 | 2
  Race: White | 18 | 42 | 22 | 82
  Race: Multiple | 1 | 0 | 0 | 1
  Race: Other | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time-Normalized Investigator-Confirmed (IC) HAE Attack Rate (Per Month) From Week 1 to Week 25
Description: The time-adjusted HAE attack rate was calculated as number of IC HAE attacks occurring from Week 1 to Week 25, divided by the number of days the participant contributed to the period multiplied by 28 days. An HAE attack was defined as an event with signs or symptoms consistent with an attack in at least 1 of the locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx).
Time Frame: Week 1 to Week 25
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: HAE attacks per month
Arm/Group | Pooled Placebo | Cohort A: Donidalorsen 80 mg | Cohort B: Donidalorsen 80 mg
Number analyzed (Participants) | 22 | 45 | 23
HAE attacks per month | 2.26 [1.657 to 3.085] | 0.44 [0.265 to 0.727] | 1.02 [0.651 to 1.594]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort A: Donidalorsen 80 mg; The Poisson regression model includes treatment groups, baseline (the run-in period HAE attack rate), the treatment-by-baseline interaction as a covariate, and the logarithm of time in every-4-week that each participant was observed from Week 1 to Week 25 used as an offset variable. Pearson chi-square scaling of standard errors was used to account for potential over dispersion; Test type: Superiority; p < 0.001, Poisson regression model; IC HAE attack rate ratio = 0.19, 95% CI 2-sided [0.107 to 0.351] — Model adjusted rate ratio from Poisson regression model
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort B: Donidalorsen 80 mg; The Poisson regression model includes treatment groups, baseline (the run-in period HAE attack rate), the treatment-by-baseline interaction as a covariate, and the logarithm of time in every-4-week that each participant was observed from Week 1 to Week 25 used as an offset variable. Pearson chi-square scaling of standard errors was used in the Poisson regression model to account for potential overdispersion; Test type: Superiority; p = 0.004, Poisson regression model; IC HAE attack rate ratio = 0.45, 95% CI 2-sided [0.261 to 0.777] — Model adjusted rate ratio from Poisson regression model

2. Secondary Outcome: Time-Normalized IC HAE Attack Rate (Per Month) From Week 5 to Week 25
Description: The time-adjusted HAE attack rate was calculated as number of IC HAE attacks occurring from Week 5 to Week 25, divided by the number of days the participant contributed to the period multiplied by 28 days. An HAE attack was defined as an event with signs or symptoms consistent with an attack in at least 1 of the locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx).
Time Frame: Week 5 to Week 25
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: HAE attacks per month
Arm/Group | Pooled Placebo | Cohort A: Donidalorsen 80 mg | Cohort B: Donidalorsen 80 mg
Number analyzed (Participants) | 22 | 45 | 23
HAE attacks per month | 2.25 [1.594 to 3.183] | 0.30 [0.151 to 0.581] | 0.90 [0.529 to 1.520]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort A: Donidalorsen 80 mg; The Poisson regression model includes treatment groups, baseline (the run-in period HAE attack rate), the treatment-by-baseline interaction as a covariate, and the logarithm of time in every-4-week that each participant was observed from Week 5 to Week 25 used as an offset variable. Pearson chi-square scaling of standard errors was used in the Poisson regression model to account for potential over dispersion; Test type: Superiority; p < 0.001, Poisson regression model; IC HAE attack rate ratio = 0.13, 95% CI 2-sided [0.062 to 0.281] — Model adjusted rate ratio from Poisson regression model
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort B: Donidalorsen 80 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.004, Poisson regression model; IC HAE attack rate ratio = 0.4, 95% CI 2-sided [0.212 to 0.748] — Model adjusted rate ratio from Poisson regression model

3. Secondary Outcome: Percentage of IC HAE Attack-Free Participants From Week 5 to Week 25
Description: An HAE attack was defined as an event with signs or symptoms consistent with an attack in at least 1 of the locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx). Percentages are rounded off to the nearest decimal.
Time Frame: Week 5 to Week 25
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Pooled Placebo | Cohort A: Donidalorsen 80 mg | Cohort B: Donidalorsen 80 mg
Number analyzed (Participants) | 22 | 45 | 23
Percentage of participants | 9.1 | 53.3 | 34.8
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort A: Donidalorsen 80 mg; Test type: Superiority; p = 0.003, Regression, Logistic; p-value was calculated based on logistic regression with baseline and the treatment-by-baseline interaction as a covariate; Odds Ratio (OR) = 11.79, 95% CI 2-sided [2.34 to 59.36]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort B: Donidalorsen 80 mg; Test type: Superiority; p = 0.240, Regression, Logistic; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 3.23, 95% CI 2-sided [0.46 to 22.85]

4. Secondary Outcome: Time-Normalized Moderate or Severe IC HAE Attack Rate (Per Month) From Week 5 to Week 25
Description: The time-adjusted HAE attack rate was calculated as number of investigator-confirmed moderate or severe HAE attacks occurring from Week 5 to Week 25, divided by the number of days the participant contributed to the period multiplied by 28 days. An HAE attack was defined as an event with signs or symptoms consistent with an attack in at least 1 of the locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx).
Time Frame: Week 5 to Week 25
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: HAE attacks per month
Arm/Group | Pooled Placebo | Cohort A: Donidalorsen 80 mg | Cohort B: Donidalorsen 80 mg
Number analyzed (Participants) | 22 | 45 | 23
HAE attacks per month | 1.15 [0.718 to 1.831] | 0.12 [0.044 to 0.351] | 0.68 [0.372 to 1.229]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort A: Donidalorsen 80 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Poisson regression model; IC HAE attack rate ratio = 0.11, 95% CI 2-sided [0.035 to 0.339] — Model adjusted rate ratio from Poisson regression model
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort B: Donidalorsen 80 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.173, Poisson regression model; IC HAE attack rate ratio = 0.59, 95% CI 2-sided [0.276 to 1.260] — Model adjusted rate ratio from Poisson regression model

5. Secondary Outcome: Number of Participants With a Clinical Response From Week 5 to Week 25
Description: Clinical response was defined as a ≥ 50%, ≥ 70%, or ≥ 90% reduction from Baseline in HAE attack rate from Week 5 to Week 25. The HAE attack rate between Week 5 and Week 25 for each participant is calculated as number of HAE attacks occurring from Week 5 to week 25 divided by the number of days the participant contributed to the period multiplied by 28 days. An HAE attack was defined as an event with signs or symptoms consistent with an attack in at least 1 of the locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx). Baseline= Run-in period which is the period from screening to the last day prior to Study Day 1.
Time Frame: Week 5 to Week 25
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | Cohort A: Donidalorsen 80 mg | Cohort B: Donidalorsen 80 mg
Number analyzed (Participants) | 22 | 45 | 23
Participants
  ≥ 50% Reduction | 6 | 42 | 19
  ≥ 70% Reduction | 4 | 37 | 15
  ≥ 90% Reduction | 2 | 28 | 11
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort A: Donidalorsen 80 mg; ≥ 50% Reduction; Test type: Superiority; p < 0.001, Regression, Logistic; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 310.35, 95% CI 2-sided [11.63 to 8279.94] — The odds ratio and its 95% confidence interval were calculated based on a logistic regression with baseline (the time-normalized run-in period attack rate) and the treatment-by-baseline interaction as a covariate
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort B: Donidalorsen 80 mg; ≥ 50% Reduction; Test type: Superiority; p < 0.001, Regression, Logistic; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 14.8, 95% CI 2-sided [3.15 to 69.41] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: Donidalorsen 80 mg; ≥ 70% Reduction; Test type: Superiority; p < 0.001, Regression, Logistic; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 34.74, 95% CI 2-sided [7.32 to 164.87] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Pooled Placebo vs Cohort B: Donidalorsen 80 mg; ≥ 70% Reduction; Test type: Superiority; p = 0.004, Regression, Logistic; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 9.17, 95% CI 2-sided [2.05 to 41.09] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Pooled Placebo vs Cohort A: Donidalorsen 80 mg; ≥ 90% Reduction; Test type: Superiority; p < 0.001, Regression, Logistic; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 17.04, 95% CI 2-sided [3.36 to 86.42] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Pooled Placebo vs Cohort B: Donidalorsen 80 mg; ≥ 90% Reduction; Test type: Superiority; p = 0.014, Regression, Logistic; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 8.7, 95% CI 2-sided [1.56 to 48.52] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: IC HAE Attack Rate Requiring Acute HAE Therapy From Week 5 to Week 25
Description: Time-adjusted HAE attack rate is calculated as number of IC HAE attacks requiring acute therapy occurring from Week 5 to Week 25, divided by number of days the participant contributed to period multiplied by 28 days. An HAE attack was defined as an event with signs or symptoms consistent with an attack in at least 1 of the locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx). HAE attacks requiring acute therapy included those attacks with following concomitant medications c1 esterase inhibitors (human and recombinant), plasma kallikrein inhibitor (human), and bradykinin antagonist.
Time Frame: Week 5 to Week 25
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: HAE attacks per month
Arm/Group | Pooled Placebo | Cohort A: Donidalorsen 80 mg | Cohort B: Donidalorsen 80 mg
Number analyzed (Participants) | 22 | 45 | 23
HAE attacks per month | 1.80 [1.232 to 2.616] | 0.15 [0.057 to 0.391] | 0.59 [0.308 to 1.146]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort A: Donidalorsen 80 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Poisson regression model; IC HAE attack rate ratio = 0.08, 95% CI 2-sided [0.030 to 0.234] — Model adjusted rate ratio from Poisson regression model
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort B: Donidalorsen 80 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.004, Poisson regression model; IC HAE attack rate ratio = 0.33, 95% CI 2-sided [0.155 to 0.706] — Model adjusted rate ratio from Poisson regression model

7. Secondary Outcome: Percentage of Participants Who Are Well Controlled on the Angioedema Control Test (AECT) at Week 25
Description: The AECT is a validated participant-reported outcome instrument to assess disease activity in participants with recurrent angioedema. The questionnaire consists of 4 questions asking about the frequency and severity of angioedema experienced in last 4 weeks. Each question has 5 response choices with total score ranging from 0 to 16. The AECT can be used to identify participants with poorly controlled disease by working with a cutoff value of greater than or equal to 10 points. Participants who score less than 10 points (0-9) in the AECT have poorly controlled disease whereas participants with well-controlled disease score 10-16 points. Percentages are rounded off to the nearest decimal.
Time Frame: Week 25
Population: The FAS included all randomized participants who received at least 1 dose of the study drug (donidalorsen or placebo). Overall number analyzed is the number of participants with data available for analysis at the specified timepoint. As pre-specified in the protocol and statistical analysis plan, for purposes of analysis, data for placebo participants from Cohort A and Cohort B was pooled for comparison to donidalorsen treated participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Pooled Placebo | Cohort A: Donidalorsen 80 mg | Cohort B: Donidalorsen 80 mg
Number analyzed (Participants) | 17 | 42 | 22
Percentage of participants | 47.1 | 92.9 | 77.3

8. Secondary Outcome: Change From Baseline in Angioedema Quality of Life (AE-QoL) Questionnaire Total Score at Week 25
Description: The AE-QoL questionnaire is a validated tool to assess symptom-specific health-related QOL impairment in participants suffering from recurrent angioedema. It is a self-administered questionnaire comprising 17 questions across 4 domains: functioning, fatigue/mood, fears/shame, and food. The responses are scored from 0 to 4 where, 0 = never, 1 = rarely, 2 = occasionally, 3 = often, 4 = very often. The AE-QoL domain scores and total score were calculated by using the following formula: (Sum score of all completed items) / (maximum sum score of all possible items) × 100. Total scores ranges from 0 to 100, with higher scores indicating greater impairment. Negative change from baseline indicates improvement. The calculated domain and total scores were not raw scores but linear transformations to a 0 to 100 scale. Baseline is defined as the score on Study Day 1.
Time Frame: Week 25
Population: The FAS included all randomized participants who received at least 1 dose of the study drug (donidalorsen or placebo). Overall number of participants analyzed is the number of participants with data available for analysis at the specified time point. As pre-specified in the protocol and statistical analysis plan, for purposes of analysis, data for placebo participants from Cohort A and Cohort B was pooled for comparison to donidalorsen treated participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pooled Placebo | Cohort A: Donidalorsen 80 mg | Cohort B: Donidalorsen 80 mg
Number analyzed (Participants) | 18 | 42 | 22
Score on a scale | -6.19 [-13.737 to 1.353] | -24.76 [-29.860 to -19.652] | -19.85 [-26.960 to -12.734]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort A: Donidalorsen 80 mg; Test type: Superiority; p < 0.001, Mixed model with repeated measures(MMRM); Treatment difference = -18.56, 95% CI 2-sided [-27.673 to -9.454]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort B: Donidalorsen 80 mg; Test type: Superiority; p = 0.010, MMRM; Treatment difference = -13.65, 95% CI 2-sided [-24.024 to -3.286]

ADVERSE EVENTS:
Time Frame: Up to Week 38
Description: The safety set included all randomized participants who received at least 1 dose of the study drug (donidalorsen or placebo). As pre-specified in the protocol and statistical analysis plan, for purposes of analysis, data for placebo participants from Cohort A and Cohort B was pooled for comparison to donidalorsen treated participants.
Arm/Group | Pooled Placebo | Cohort A: Donidalorsen 80 mg | Cohort B: Donidalorsen 80 mg
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/45 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/45 | 0/23
Other Adverse Events (participants affected / at risk) | 15/22 | 22/45 | 13/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=22) | Cohort A: Donidalorsen 80 mg (N=45) | Cohort B: Donidalorsen 80 mg (N=23)
Limb Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=22) | Cohort A: Donidalorsen 80 mg (N=45) | Cohort B: Donidalorsen 80 mg (N=23)
Headache (Nervous system disorders) | 4 | 7 | 2
Injection Site Erythema (General disorders) | 0 | 6 | 1
Nasopharyngitis (Infections and infestations) | 5 | 6 | 3
Influenza (Infections and infestations) | 2 | 4 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 4 | 3
Urinary Tract Infection (Infections and infestations) | 0 | 4 | 2
Injection Site Discolouration (General disorders) | 0 | 3 | 1
Injection Site Pruritus (General disorders) | 0 | 3 | 0
Injection Site Pain (General disorders) | 0 | 3 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 3 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 1 | 0
Covid-19 (Infections and infestations) | 3 | 1 | 1
Gastroenteritis (Infections and infestations) | 2 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 3 | 0 | 1
Oral Herpes (Infections and infestations) | 0 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 3
Sinusitis (Infections and infestations) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between Principal Investigators and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT05139810/Prot_SAP_000.pdf